CLINICAL TRIAL: NCT04893447
Title: Comparing the Effectiveness of Safety Planning Plus Follow-Up From a Suicide Prevention Hotline (SPI+) vs Safety Planning Plus Caring Contacts (SP+CC) Among Adults and Adolescents at Risk for Suicide in Primary Care or Emergency Departments
Brief Title: Suicide Prevention Among Recipients of Care
Acronym: SPARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Health System, Boise, Idaho (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Idaho Crisis & Suicide Hotline (Other); University of Washington (Other); Columbia University (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Anna Radin, Applied Research Scientist, St. Luke's Health System, Boise, Idaho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-0026
Record Dates: First submitted 2021-04-28; First posted 2021-05-19 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Suicide; Suicide, Attempted; Suicidal Ideation; Social Support; Secondary Prevention; Patient Care Planning; Outpatients; Outpatient Clinics, Hospital; Mental Health Services; Mental Health; Mental Disorder; Loneliness; Emergency Service, Hospital; Depressive Disorder; Depression; Continuity of Patient Care; Ambulatory Care; Adolescent; Adult; Crisis Intervention
Keywords: Brief Interventions; Caring Contacts; Care Transitions; Follow-up; Emergency Department; Primary Care; Safety Planning Intervention; Safety Plan; Suicide; Suicide Prevention; Adult; Adolescent; Brief Contact Intervention
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation; Psychological Well-Being; Mental Disorders; Emergencies; Depressive Disorder; Depression; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Individual-level randomization to one of two treatment arms
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPI+: Safety Planning Intervention plus structured phone-based follow-up (Experimental): The Safety Planning Intervention (SPI+) includes safety planning (moderate or high risk for suicide) or connection & support planning (low risk for suicide) at the clinic or ED, plus a structured telephone-based intervention from a suicide prevention hotline
  Interventions: Behavioral: SPI+
- Caring Contacts: Safety Planning Intervention plus Caring Contacts (SP+CC) (Experimental): SP+CC will include safety planning (moderate or high risk for suicide) or connection & support planning (low risk for suicide) at the clinic or ED, plus caring text messages or emails from a suicide prevention hotline.
  Interventions: Behavioral: SP+CC (Caring Contacts)

INTERVENTIONS:
Behavioral: SPI+ — Suicide prevention hotline follow-up specialists will call participants to (1) conduct a brief suicide risk assessment; (2) review and discuss the participant's connection and support plan or safety plan; and (3) provide referrals to social services or other support with treatment engagement, if indicated. Participants will receive at least one and optional additional phone calls, generally delivered according to the following schedule: days 3, 7, 14, 30, 60, 90. Modifications may be made to the schedule due to weekends, holidays, or participant availability, and additional calls may be scheduled as desired by the participant. The follow-up will stop once the participant is successfully engaged in outpatient treatment or does not desire further follow-up support.
  Other Names: phone-based follow-up, brief contact intervention
  Arms: SPI+: Safety Planning Intervention plus structured phone-based follow-up
Behavioral: SP+CC (Caring Contacts) — SP+CC follow-up includes one phone conversation with a suicide prevention hotline follow-up specialist and a series of personalized caring messages sent over the course of 12 months via text or email (based on participant preference). Caring contacts will generally be sent according to the following schedule: 3 in the first week, 6 weekly, 6 bi-weekly, 4 monthly; 2 bi-monthly, and one each for the participant's birthday, Thanksgiving, Christmas, and New Year's (total of 25 over 12 months). Slight variation in the schedule is allowed. There is no expectation that participants respond to the text messages; if they do, follow-up specialists reply to any incoming texts. Replies are individually-tailored and caring.
  Other Names: Brief contact intervention, text-based follow-up, email follow-up
  Arms: Caring Contacts: Safety Planning Intervention plus Caring Contacts (SP+CC)

SUMMARY:
Randomized controlled trial to determine the best brief suicide prevention intervention for adults and adolescents who screen positive for suicidal ideation or behavior in emergency departments or primary care clinics.

Aim 1: Compare the effectiveness of two brief suicide prevention interventions (safety planning intervention plus structured phone-based follow-up from a suicide prevention hotline (SPI+), versus safety planning intervention plus caring contacts (CC)) to (a) reduce suicidal ideation and behavior, (b) reduce loneliness, (c) reduce return to care for suicidality, and (d) increase uptake of outpatient mental healthcare services over 12 months among adult and adolescent patients screening positive for suicide in emergency departments (EDs) and primary care clinics.

Aim 2: Assess the acceptability of connection and support planning and the safety planning intervention, with or without follow-up among providers and clinical staff in EDs and primary care clinics.

Aim 3: Assess the acceptability of SPI+ and SP+CC among adult and adolescent patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient at St. Luke's Health System Emergency Department or Primary Care Clinic
* 12-17 years old (adolescents) or 18+ years old (adults)
* Screened positive for suicide risk on C-SSRS (any response of "yes") during current visit, or current visit is related to a suicide attempt
* Access to a phone for the duration of the study with the ability to receive calls
* The ability to send and receive email messages (required) and text messages (optional)
* English or Spanish speaking and reading

Exclusion Criteria:

* Unable or unwilling to provide informed consent to participate
* Inappropriate for study participation based on the clinical judgment of provider

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1520 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Suicidal Ideation & Behavior; measured using the Columbia Suicide Severity Rating Scale (C-SSRS) since-last-contact screener (self-assessment) | 6 months
  6-item questionnaire with yes/no response options. Scores range from 0 (no risk) to 6 (high risk)

SECONDARY OUTCOMES:
Loneliness; measured using the NIH Toolbox Emotion Batteries Loneliness Scale | 6 months
  5-item questionnaire with Likert scale response options (1=never, 5=always). Scores range from 5 (no loneliness) to 25 (high levels of loneliness).
Loneliness; measured using the NIH Toolbox Emotion Batteries Loneliness Scale | 12 months
  5-item questionnaire with Likert scale response options (1=never, 5=always). Scores range from 5 (no loneliness) to 25 (high levels of loneliness).
Utilization of Emergency Department for Suicidality | 6 months
  Measured through self-report
Utilization of Emergency Department for Suicidality | 12 months
  Measured through self-report
Attendance at Outpatient Behavioral Health Appointments | 6 months
  Measured through self-report
Attendance at Outpatient Behavioral Health Appointments | 12 months
  Measured through self-report
Suicidal Ideation & Behavior; measured using the Columbia Suicide Severity Rating Scale (C-SSRS) since-last-contact screener (self-assessment) | 12 months
  6-item questionnaire with yes/no response options. Scores range from 0 (no risk) to 6 (high risk)

CONTACTS AND LOCATIONS:
Overall Officials: Anna K Radin, DrPH, MPH, Principal Investigator — St. Luke's Health System
Locations (1):
- St. Luke's Health System, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: Yes
After publication of the final research report, de-identified data may be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data are estimated to become available in 2026.
Access Criteria: A data access committee will review and make decisions on all requests to access data.

DOCUMENTS (2):
  • Study Protocol (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT04893447/Prot_000.pdf
  • Informed Consent Form (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT04893447/ICF_001.pdf